CLINICAL TRIAL: NCT04378062
Title: Pain After Proximal Digital Amputation Prevention
Acronym: PAPDAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate enrollment
Sponsor: Indiana University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Principal Investigator, Joshua Adkinson, Assistant Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1907889836
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pain; Amputation Neuroma; Amputation
Keywords: Pain; Amputation Neuroma; Finger Amputation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traction Neurectomy (Active Comparator): Traction neurectomy - of digital sensory nerves at the time of amputation.
  Interventions: Procedure: Digital nerve procedure
- Targeted Muscle Reinnervation (Experimental): Targeted Muscle Reinnervation - of digital sensory nerves at the time of amputation
  Interventions: Procedure: Digital nerve procedure
- Regenerative Peripheral Nerve Interface (Experimental): Regenerative Peripheral Nerve Interface - of digital sensory nerves at the time of amputation
  Interventions: Procedure: Digital nerve procedure

INTERVENTIONS:
Procedure: Digital nerve procedure — The type of procedure performed on the digital nerve at the time of amputation

SUMMARY:
Finger amputations are common and may be complicated by debilitating nerve pain. This study seeks to determine if nerve pain after digital amputation can be more effectively prevented with either of two new surgical techniques-targeted muscle reinnervation (TMR) or regenerative peripheral nerve interfaces (RPNI)-compared to standard treatment by traction neurectomy (TN).

DETAILED DESCRIPTION:
Patients who require proximal amputations will have the opportunity to enroll in the study, will be randomized intraoperatively to receiving one of the aforementioned treatments, and will be followed at 3 and 6 month for outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring single finger amputations at the level of the proximal interphalangeal joint or proximal (i.e., closer to the body than this joint).
* Patients have the capacity to complete the informed consent process

Exclusion Criteria:

* Patients less than 18 years of age, prisoner, or other vulnerable population
* Patients with significant concomitant ipsilateral extremity injuries that would confound study
* Patients requiring emergent, staged (guillotine-type) amputations of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
bMHQ | 3 months postop minus preop; 6 months postop minus preop
  Breif Michigan Hand Questionnaire Score difference

SECONDARY OUTCOMES:
NPS | 3 months postop minus preop; 6 months postop minus preop
  Numerical Pain Score difference
Grip strength | 3 months postop minus preop; 6 months postop minus preop
  Grip strength score difference

OTHER OUTCOMES:
Tinel's sign | Tinel's sign at 3 months; Tinel's sign at 6 months
  Tinel's sign at amputation site

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Adkinson, MD, Principal Investigator — Indiana University; Scott N Loewenstein, MD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No